CLINICAL TRIAL: NCT02402556
Title: Implementation and Impact Evaluation of the Mother and Child Education Program (MOCEP) Among Children and Families in Palestinian Refugee Camps in Beirut, Lebanon
Brief Title: Mother and Child Education Program in Palestinian Refugee Camps
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 1403013605
Record Dates: First submitted 2015-03-25; First posted 2015-03-30 (Estimated); Last update posted 2016-12-02 (Estimated); Status verified 2016-12

CONDITIONS: Parenting

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MOCEP (Experimental): MOCEP is implemented over a period of 25 weeks, through weekly group meetings that last approximately three hours.
  Interventions: Behavioral: MOCEP
- Waitlist Control Group (Active Comparator): For ethical reasons, no one recruited will be excluded from the opportunity to benefit from the intervention. MOCEP group will be the primary intervention group and the second group will act as the wait-listed control group. Although the families in the wait-listed control group will start out as a control group (not receiving the intervention), they will have the opportunity to participate in the intervention in a later round of implementation, after the intervention group has completed the program.
  Interventions: Behavioral: MOCEP

INTERVENTIONS:
Behavioral: MOCEP — Through parent support and an evidence-based curriculum, MOCEP uses education to reduce risk factors that hinder children's health and wellbeing.

SUMMARY:
The purpose of the Mother Child Education Program (MOCEP)-a group-based early childhood development parenting education program-is to provide school-readiness and parenting skills to mothers of young children who do not have access to preschool education services. The MOCEP intervention also provides a setting in which caregivers can model pro-social behaviors and practice conflict resolution techniques directly with young children.

DETAILED DESCRIPTION:
The purpose of the evaluation study is to rigorously evaluate the impact of MOCEP on child and parent outcomes among Palestinian refugees in Beirut, Lebanon. This evaluation employs an innovative, mixed-methods bio-behavioral approach to investigate the associations among social contexts; maternal, child and family functioning; and reduction in violence through the promotion of harmonious family relationships. The results of this study have implications for improving the lives of and reducing violence for the hundreds of thousands of families with young children living in fragile contexts. We hypothesize that when MOCEP is implemented with fidelity (i.e., delivered as intended by design), participating families will experience reduced violence in their homes and have better individual and intra-family outcomes than families who do not participate in the program.

ELIGIBILITY:
Inclusion Criteria:

1. Child must be between 3 and 6 years of age (children age 7 may be accepted under special circumstances)
2. Mother must be able to read and write in Arabic (although skills may not be well-developed)
3. Mothers must commit to participate in the 25-week MOCEP Intervention program

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 106 (Actual)
Dates: Start 2014-05; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Disciplinary Style Questionnaire | 25 weeks
  Parent report measure of parental disciplinary style assesses the frequency with which parents engage in seven forms of discipline when dealing with children's undesirable behavior
Better Parenting Questionnaire | 25 weeks
  11 Item questionnaire that measures parental knowledge, attitudes and practices regarding education and learning, child development and discipline / child rearing.

SECONDARY OUTCOMES:
Socio-Emotional Status: Strengths and Difficulties Questionnaire (child assessment) | 25 weeks
  Parent report measure assesses children's emotional and conduct problems, hyperactivity, and peer relations.
Parental Stress Index | 25 weeks
  Assessment of maternal stress
Duke Social Support Index | 25 weeks
  Addresses social support in two domains: social interaction and subjective support

CONTACTS AND LOCATIONS:
Overall Officials: James Leckman, MD, Principal Investigator — Yale University
Locations (3):
- Lebanon (3):
  - Bourj el-Barajneh refugee camp, Beirut
  - Charila, Beirut
  - Mar Elias Refugee Camp, Beirut

REFERENCES:
- [Derived] Ponguta LA, Issa G, Aoudeh L, Maalouf C, Hein SD, Zonderman AL, Katsovich L, Khoshnood K, Bick J, Awar A, Nourallah S, Householder S, Moore CC, Salah R, Britto PR, Leckman JF. Effects of the Mother-Child Education Program on Parenting Stress and Disciplinary Practices Among Refugee and Other Marginalized Communities in Lebanon: A Pilot Randomized Controlled Trial. J Am Acad Child Adolesc Psychiatry. 2020 Jun;59(6):727-738. doi: 10.1016/j.jaac.2019.12.010. Epub 2020 Jan 31. PMID 32014538